CLINICAL TRIAL: NCT00648089
Title: ErythroPOietin in Myocardial Infarction
Brief Title: EPOMI Study: ErythroPOietin in Myocardial Infarction
Acronym: EPOMI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Collaborators: Fédération Française de Cardiologie (Other); Société Française de Cardiologie (Other)
Responsible Party: Fabrice PRUNIER, MD, PhD, University Hospital, Angers
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHRC 2007-03
Record Dates: First submitted 2008-03-27; First posted 2008-04-01 (Estimated); Last update posted 2011-01-31 (Estimated); Status verified 2011-01

CONDITIONS: Myocardial Infarction
Keywords: Acute ST Elevation Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: EPO
- 2 (No Intervention)

INTERVENTIONS:
Drug: EPO — Single Injection of 1000 U/kg Erythropoietin beta IV immediately after primary PCI
  Arms: 1

SUMMARY:
EPOMI is a randomized, open-label, parallel phase II clinical study that will evaluate the effects of a single erythropoietin administration on infarct size and cardiac remodeling in patients with acute myocardial infarction. Eligible patients will be randomly assigned to receive conventional therapy and single infusion of 1000U/kg of epoetin beta or conventional therapy alone. Infarct size and cardiac remodeling parameters will be assessed by cardiac magnetic resonance imaging (MRI) within 3-7 days of the randomization and repeated 3 months later.

ELIGIBILITY:
Inclusion Criteria:

* ST-Segment elevation myocardial infarction <6h
* Infarct related artery : proximal circumflex artery , proximal and mid left anterior descending artery, 1st segment of the right coronary artery
* TIMI 0 or 1 before angioplasty
* Successful PCI defined by residual stenosis < 50% and TIMI 2 or 3 flow grade
* Body weight : [50-110] kg
* Informed, written consent

Exclusion Criteria:

* Age < 18
* Pregnant, or parturient or breast-feeding women;
* Sexually active women without efficient contraception;
* Inability to fully cooperate with the study protocol
* Pre-treatment with fibrinolysis ;
* Previous Q-wave myocardial infarction or previous aorto-coronary bypass;
* History of deep vein thrombosis or pulmonary embolism;
* Contraindication to aspirin or clopidogrel ;
* Cardiogenic shock ;
* Cardiac resuscitated before angioplasty ;
* Past or active erythropoietin therapy;
* Contraindications to erythropoietin therapy: uncontrolled hypertension, known hypersensitivity to benzoic acid, chronic liver insufficiency, hemoglobin> 16g / l, thrombocytosis, refractory anemia with excess of blasts;
* Renal insufficiency (creatinine clearance <30ml/mn.);
* Active Malignancies
* Any contraindications to magnetic resonance imaging: pacemaker and automatic cardiac defibrillator, hearing aid, neurostimulator, infusion pump etc metallic splinters in the eye, ferromagnetic haemostatic clips in the central nervous system cochlear implants, claustrophobia;
* Allergy to gadolinium ;
* Patient refusal / patient not having provided written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2008-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Changes in infarct size as assessed by magnetic resonance imaging 3 months after administration of study medication | within 3-7 days of administration of study medication

SECONDARY OUTCOMES:
End-systolic volume, end-diastolic volume, ejection fraction | within 3-7 days of administration of study medication, and 3 months later
Changes in hemoglobin, platelets, reticulocytes blood count | during the first 10 days following study medication administration
Occurrence of major cardiac event or venous thrombotic events | within 12 months following administration of study medication

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice PRUNIER, MD, PhD, Principal Investigator — University Hospital, Angers
Locations (2):
- France (2):
  - CHU Angers, Angers
  - Fabrice PRUNIER, MD, PhD,, Angers

REFERENCES:
- [Derived] Prunier F, Biere L, Gilard M, Boschat J, Mouquet F, Bauchart JJ, Charbonnier B, Genee O, Guerin P, Warin-Fresse K, Durand E, Lafont A, Christiaens L, Abi-Khalil W, Delepine S, Benard T, Furber A. Single high-dose erythropoietin administration immediately after reperfusion in patients with ST-segment elevation myocardial infarction: results of the erythropoietin in myocardial infarction trial. Am Heart J. 2012 Feb;163(2):200-7.e1. doi: 10.1016/j.ahj.2011.11.005. PMID 22305837